CLINICAL TRIAL: NCT05815238
Title: Changes in Foot Posture With Age: Functional and Balance Effects
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, Principal Investigator, Istanbul Medipol University Hospital
Other Study IDs: Foot Posture Index
Record Dates: First submitted 2023-04-04; First posted 2023-04-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Foot Posture Index Score
Keywords: balance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Young Adult: 20-35
- Mild Adults: 35-50
- Older Adults: 50-65

SUMMARY:
The foot is a terminal joint that opposes external resistance in the lower kinetic chain. It plays a primary role in weight transfer and ground response between the body and the ground. It plays a role in maintaining an upright posture, lowering the gravitational line against a narrow support surface during walking, providing stability and absorbing the shocks that occur during daily life activities.

Foot problems are common worldwide. These problems affect people negatively by giving symptoms during activities of daily living.

DETAILED DESCRIPTION:
There is not much data on whether these changes are related to age or not. Deformities, kinetic chain disorders, and other problems that affect balance are likely to increase with age. For this reason, in our study, the relationship between foot posture and functional-balance was examined on the basis of age groups.

Body balance may be impaired by deficiencies in the strength and mechanical stability of any joint or structure along the lower extremity kinetic chain, or by decreased afferent feedback. It is necessary to know the foot posture and biomechanics about the causes of injury and susceptibility to injury during activities of daily living and sports.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 20 - 65,
* Volunteer.

Exclusion Criteria:

* Having a musculoskeletal or neuromuscular disease that limits mobility,
* Presence of lower extremity sequelae,

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals who will participate in the study will be reached via social media, whatsapp and message.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-09-26 (Actual)

PRIMARY OUTCOMES:
Foot Function Index | 1 day
  The foot function index was developed and widely used to measure the effects of foot pathologies on pain, disability and activity limitation.
  Foot function index; It consists of 23 items in 3 groups as pain, disability and activity limitation. While the pain and disability section consists of 9 questions, the activity limitation consists of 5 questions.
  The patients answer all the items considering their foot condition one week ago. The score of each section and the total score are calculated and we divide by the sum of the maximum scores of the items and multiply by 100.
Foot Posture Index | 1 day
  Foot Posture consists of palpation of 6 regions.
  1. Talus head palpation
  2. Curvature above and below the lateral malleolus
  3. Inversion and eversion of os calcaneus
  4. Protrusion in the talonavicular joint area
  5. Harmony of the medial longitudinal arch
  6. Abduction and adduction of the forefoot section relative to the hindfoot section.
  Each criterion is evaluated between -2 and +2 and this result is noted. Positive values indicate pronation, negative values indicate supination.
Single Leg Jump Test (TBS) | 1 day
  TBS test will be applied to evaluate the lower extremity functional performances of healthy individuals. While individuals are standing on one leg, the other leg is asked to jump forward with the knee bent and the point where the fingertip touches is marked. The jump distance is measured and the test is repeated 3 times and the average result is obtained. In our study, the single leg jump test will be used for both legs.
Y Balance Test | 1 day
  The leg lengths of all individuals are measured bilaterally. While measuring, individuals are asked to lie in their anterior, posteromedial and posterolateral directions. Each of the participants is informed before the measurement. Measurements were made in both legs and will be repeated 3 times. When calculating the total score, the values in centimeters of the 3 directions are added. Divide by the product of the length of the leg by 3 and multiply the result by 100 to reach the percentile.

CONTACTS AND LOCATIONS:
Locations (1):
- HAZAL genç, Istanbul, Turkey (Türkiye)